CLINICAL TRIAL: NCT03252496
Title: Combined Colloids And Crystalloids Versus Crystalloids in Women With Preeclampsia Undergoing Cesarean Delivery Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: Combined Colloids And Crystalloids Versus Crystalloids in Women With Preeclampsia Undergoing Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Lecturer, Department of anesthesia and surgical intensive care, Primary investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R/17.06.79
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Pre-Eclampsia; Cesarean Section
MeSH Terms: conditions — Pre-Eclampsia | interventions — Anesthesia, Spinal; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination (Experimental): 250 mL colloid over 5 minutes followed by 500 mL crystalloid over 55 minutes then 250 mL colloid over 60 minutes. Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 μg). Ultrasound assessment of the Inferior vena cava diameter. Intravenous ephedrine and intravenous syntocinon will be administered.
  Interventions: Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl; Procedure: Cesarean Delivery; Radiation: Ultrasound Assessment of the Inferior Vena Cava; Drug: 250 mL Colloid over 5 minutes; Drug: 500 mL Crystalloid over 55 minutes; Drug: 250 mL Colloid over 60 minutes; Drug: Intravenous Ephedrine; Drug: Intravenous Syntocinon
- Crystalloid (Active Comparator): 250 mL crystalloid over 5 minutes followed by 500 mL crystalloid over 55 minutes then 250 mL crystalloid over 60 minutes. Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 μg). Ultrasound assessment of the Inferior vena cava diameter. Intravenous ephedrine and intravenous syntocinon will be administered.
  Interventions: Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl; Procedure: Cesarean Delivery; Radiation: Ultrasound Assessment of the Inferior Vena Cava; Drug: 250 mL Crystalloid over 5 minutes; Drug: 500 mL Crystalloid over 55 minutes; Drug: 250 mL Crystalloid over 60 minutes; Drug: Intravenous Ephedrine; Drug: Intravenous Syntocinon

INTERVENTIONS:
Procedure: Spinal Anesthesia — Performed at the L3-L4 or L4-L5 interspace using 27- or 25-gauge spinal needle
Drug: Intrathecal Bupivacaine — Bupivacaine 12.5 mg (2.5 mL 0.5%) will be administered in the subarachnoid space
Drug: Intrathecal Fentanyl — Fentanyl 15 μg will be administered in the subarachnoid space
Procedure: Cesarean Delivery — Lower segment cesarean section using the Pfannenstiel incision
Radiation: Ultrasound Assessment of the Inferior Vena Cava — The inferior vena cava largest and smallest diameters will be measured proximal to the opening of the hepatic veins in the longitudinal axis with the M-mode using a 8-2 MHz curved array ultrasound probe placed longitudinally in the subcostal region
Drug: 250 mL Colloid over 5 minutes — 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride (voluven®) 250 mL will be administered over 5 minutes starting immediately after intrathecal injection
  Arms: Combination
Drug: 250 mL Crystalloid over 5 minutes — Ringer acetate 250 mL will be administered over 5 minutes starting immediately after intrathecal injection
  Arms: Crystalloid
Drug: 500 mL Crystalloid over 55 minutes — Ringer acetate 500 mL will be administered over 55 minutes following colloid or crystalloid administration
Drug: 250 mL Colloid over 60 minutes — After 60 minutes of intrathecal injection, 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride (voluven®) 250 mL will be administered over 60 minutes
  Arms: Combination
Drug: 250 mL Crystalloid over 60 minutes — After 60 minutes of intrathecal injection, Ringer acetate 250 mL will be administered over 60 minutes
  Arms: Crystalloid
Drug: Intravenous Ephedrine — Intravenous ephedrine 3, 5, and 10 mg will be administered when Systolic blood pressure decreases below 120, 110, and 90 mmHg, respectively.
Drug: Intravenous Syntocinon — Immediately after delivery, syntocinon 10 IU will be added to the running crystalloid solution

SUMMARY:
This study will compare between combination of colloids/crystalloids and crystalloids in women with preeclampsia undergoing elective cesarean delivery under spinal anesthesia

DETAILED DESCRIPTION:
This randomized, controlled, double blind study will be conducted on women with preeclampsia with singleton pregnancy undergoing elective cesarean delivery under spinal anesthesia. Immediately, after spinal anesthesia administration, patients will receive either 250 mL colloid over 5 minutes followed by 500 mL crystalloid over 55 minutes then 250 mL colloid over 60 minutes (Combination group) or 250 mL crystalloid over 5 minutes followed by 500 mL over 55 minutes then 250 mL over 60 minutes (Crystalloid group). The studied maternal outcomes will be the urine output, ephedrine requirement, incidence of hypotension, inferior vena cava diameters, nausea/vomiting and bradycardia. Neonatal Apgar scores will be recorded at 1 and 5 minutes post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia: Blood Pressure ≥140/90 mmHg after 20 weeks' gestation and proteinuria ≥300 mg/24 hours or 1+ on urine dipstick
* Singleton pregnancy
* Elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Height <150 cm
* Weight <60 kg
* Body mass index ≥45 kg/m2
* Women presenting in labor
* Contraindications to spinal anesthesia (increased intracranial pressure or local skin infection)
* Diabetes mellitus, cardiovascular, cerebrovascular, or renal disease
* Preoperative administration of intravenous hydralazine or magnesium sulphate
* Hemoglobin <10 gm/dL
* International Normalized Ratio >1.3
* Platelet count <100,000 /mm3
* Preoperative serum creatinine >1.1 mg/dL

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Total urine output at 2 hours post-spinal | 2 hours after intrathecal injection

SECONDARY OUTCOMES:
Urine output at 1 hour post-spinal | 1 hour after intrathecal injection
Incidence of oliguria | 2 hours after intrathecal injection
  Total urine output at 2 hours post-spinal <60 mL
Total ephedrine dose | Intraoperative
Pre-delivery ephedrine dose | From intrathecal injection until delivery
Number of patients requiring ephedrine | Intraoperative
Number of patients requiring ephedrine pre-delivery | From intrathecal injection until delivery
Incidence of nausea and/or vomiting | Intraoperative
Incidence of bradycardia | Intraoperative
  Heart rate <50 beats/minute
Maximum and minimum inferior vena cava diameters | Baseline, at 5 minutes post-spinal, immediately after delivery of the fetus, and at 1 and 2 hours post-spinal
Inferior vena cava collapsibility index | Baseline, at 5 minutes post-spinal, immediately after delivery of the fetus, and at 1 and 2 hours post-spinal
Neonatal Apgar score | At 1 and 5 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Tawfik, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No